CLINICAL TRIAL: NCT03817164
Title: Multicenter, Randomized, Double-Blind, Sham-Controlled, Efficacy and Safety Study of Autonomic Nerve Modulation (ANM) in Subjects With Moderate Plaque Psoriasis
Brief Title: Efficacy and Safety Study of Autonomic Nerve Modulation (ANM) in Subjects With Moderate Plaque Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thync Global, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THY-004
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Active Comparator): Active stimulation pulsed current delivered over 15 minutes.
  Interventions: Device: Autonomic Nerve Modulation - Active
- Control Treatment (Sham Comparator): Active stimulation pulsed current (alternative frequency) delivered over 15 minutes.
  Interventions: Device: Autonomic Nerve Modulation - Control

INTERVENTIONS:
Device: Autonomic Nerve Modulation - Active — Thync ANM is a portable, battery-powered, electrical neuromodulation device connected to single-use gel electrode pads that are applied to the base of the neck.
  Arms: Active Treatment
Device: Autonomic Nerve Modulation - Control — Thync ANM is a portable, battery-powered, electrical neuromodulation device connected to single-use gel electrode pads that are applied to the base of the neck.
  Arms: Control Treatment

SUMMARY:
This is a 16-week, prospective, multicenter, double-blind, controlled, randomized study assessing change in psoriasis severity and level of stress in patients with moderate psoriasis treated with ANM. Psoriasis severity and stress levels will be measured at Weeks 0, 2, 8, 12, and 16.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female of any race, 18 years of age or older. This study has no pregnancy restrictions.
2. BSA* <10% (excluding palms, soles, intertriginous and inverse areas).
3. sPGA* ≥3 (NOTE: sPGA score will be averaged across all lesions as opposed to grading target lesions).
4. BSA x sPGA ≥12.
5. Subject diagnosed with chronic plaque psoriasis at least 6 months prior to screening.
6. Treatment-naïve of prohibited biological immunomodulating agents at the time of screening, or decided to stop treatment with the biologic before screening for the study.
7. Be able to follow study instructions and likely to complete all required visits.
8. Sign the IRB-approved ICF (which includes HIPAA).

Exclusion Criteria:

1. Non-plaque psoriasis (erythrodermic or pustular), guttate, inverse psoriatic arthritis, or drug-induced psoriasis.
2. Subjects with plaque psoriasis on palms and soles at enrolment.
3. Subjects with plaque psoriasis on the back of the neck that would interfere with device placement.
4. Evidence of skin conditions other than psoriasis that would interfere with study-related evaluations of psoriasis.
5. Other than psoriasis, history of any clinically significant (as determined by Investigator) or other major uncontrolled disease.
6. Psoriasis flare or rebound within 4 weeks of Visit 1 or spontaneously improving or rapidly deteriorating plaque psoriasis during that same time period, as determined by investigator.
7. Use of prohibited medications within the following washout periods:

   * Biological immunomodulating agents within the prior 12 weeks: etanercept (Enbrel), adalimumab (Humira), infliximab (Remicade), certolizumab pegol (Cimzia), ixekizumab (Taltz)
   * Biological immunomodulating agents within the prior 24 weeks: ustekinumab (Stelara), secukinumab (Cosentyx), guselkumba (Tremfaya)
   * Oral drugs within the prior 4 weeks: apremilast, methotrexate, cyclosporine, corticosteroids
   * Oral drugs within the prior 12 weeks: acitretin
   * Photochemotherapy (PUVA) within the prior 4 weeks
   * Phototherapy (UVA/UVB) within the prior 2 weeks
   * Topical treatment likely to impact signs and symptoms of psoriasis (e.g., corticosteroids, vitamin D analogues, retinoids, calcineurin inhibitors, salicylic acid, lactic acid, tar, urea, etc.) within the prior 2 weeks
8. Prolonged sun exposure or use of tanning booths or other source of UV radiation.
9. Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results or compliance of the subject and, in the opinion of the PI, would make the subject inappropriate for entry into this study.
10. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
11. Exposure to any other investigational drug/device within 30 days prior to study entry.
12. Subjects with a pacemaker, or any type of metal implant in the neck (i.e., T5 and above).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
BSA x sPGA average percent change from Baseline | Week 16
  Body Surface Area x Static Physician Global Assessment

SECONDARY OUTCOMES:
sPGA change from Baseline | Week 16
  Static Physician Global Assessment
BSA change from Baseline | Week 16
  Body Surface Area
Mean PASI change from Baseline | Week 16
  Psoriasis Area and Severity Index
PASI 50 | Week 16
  Psoriasis Area and Severity Index - 50% reduction
PASI 75 | Week 16
  Psoriasis Area and Severity Index - 75% reduction
PSSI change from Baseline | Week 16
  Psoriasis Scalp Severity Index
QVAS change from Baseline | Week 16
  Stress Level Quantified Visual Analogue Scale
DLQI change from Baseline | Week 16
  Dermatology Life Quality Index
PQOL-12 change from Baseline | Week 16
  Psoriasis Quality of Life - 12 Item
HADS change from Baseline | Week 16
  Hospital Anxiety and Depression Scale
Pruritus NRS change from Baseline | Week 16
  Pruritus Numerical Rating Scale
Pruritus NRS responder rate (i.e., proportion of subjects achieving a ≥4-point improvement) | Week 16
  Pruritus Numerical Rating Scale
TSQM | Week 16
  Treatment Satisfaction Questionnaire for Medication

OTHER OUTCOMES:
sPGA responder rate (i.e., proportion of subjects achieving sPGA 0 or 1) | Week 16
  Static Physician Global Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Fremont, California, United States

IPD SHARING:
Plan to Share IPD: No